CLINICAL TRIAL: NCT01212575
Title: A Retrospective, Non-interventional Study to Evaluate the Use of Seroquel XR and Seroquel IR in the Clinical Practice of Outpatients With Schizophrenia
Brief Title: A Retrospective NIS to Evaluate the Use of Seroquel XR and IR in the Clinical Practice of Outpatients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Eva Dencker Vansvik, Marketing Company Medical Director (MC MD), AstraZeneca
Other Study IDs: NIS-NDK-SER-2010/2
Record Dates: First submitted 2010-09-27; First posted 2010-09-30 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia
Keywords: Mental disorder; Antipsychotic treatment
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 300 patients: Female or male aged 18-65 years with a diagnosis of schizophrenia having received at least one dose of Seroquel XR or Seroquel IR during January - March 2010

SUMMARY:
The primary objective of this non-interventional study is to investigate how Seroquel XR and Seroquel IR are used in the clinical practice of outpatients with schizophrenia. This will be done by a retrospective review of medical records to evaluate patients treated with Seroquel XR or Seroquel IR as primary antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of schizophrenia from a district psychiatric clinic in Denmark
* Patients who have received at least one dose of Seroquel XR or Seroquel IR during January - March 2010

Exclusion Criteria:

* Patients already participating in a clinical study during the study-period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of schizophrenia who are registered at an outpatient district psychiatric clinic
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
How Seroquel XR and Seroquel IR are used in the clinical practice of outpatients with schizophrenia | Month 1
How Seroquel XR and Seroquel IR are used in the clinical practice of outpatients with schizophrenia | Month 2
How Seroquel XR and Seroquel IR are used in the clinical practice of outpatients with schizophrenia | Month 3

SECONDARY OUTCOMES:
Co-morbidities of patients with schizophrenia receiving Seroquel XR and IR | Month 1
Co-morbidities of patients with schizophrenia receiving Seroquel XR and IR | Month 2
Co-morbidities of patients with schizophrenia receiving Seroquel XR and IR | Month 3
Whether Seroquel XR and Seroquel IR are used to treat different types of outpatients with schizophrenia by evaluation of patient characteristics | Month 1
Whether Seroquel XR and Seroquel IR are used to treat different types of outpatients with schizophrenia by evaluation of patient characteristics | Month 2
Whether Seroquel XR and Seroquel IR are used to treat different types of outpatients with schizophrenia by evaluation of patient characteristics | Month 3
The treatment sequence of Seroquel XR and Seroquel IR in the clinical practice of patients with schizophrenia by evaluation of duration, dosage, reason for treatment, and, if applicable, reason for change, with Seroquel XR and Seroquel IR | Month 1
The treatment sequence of Seroquel XR and Seroquel IR in the clinical practice of patients with schizophrenia by evaluation of duration, dosage, reason for treatment, and, if applicable, reason for change, with Seroquel XR and Seroquel IR | Month 2
The treatment sequence of Seroquel XR and Seroquel IR in the clinical practice of patients with schizophrenia by evaluation of duration, dosage, reason for treatment, and, if applicable, reason for change, with Seroquel XR and Seroquel IR | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dencker Vansvik, Study Director — AstraZeneca Nordic-Södertälje, Sweden; Charlotte Emborg, Principal Investigator — Skovager 2, Risskov, Denmark
Locations (13):
- Denmark (13):
  - Research Site, Aabenraa, Aabenraa
  - Research Site, Aarhus, Arhus
  - Research Site, Arhus N, Arhus
  - Research Site, Arhus S, Arhus
  - Research Site, Ballerup Municipality, Ballerup
  - Research Site, Cph NV, Cph
  - Research Site, Cph N, Cph
  - Research Site, Esbjerg, Esbjerg
  - Research Site, Haderslev, Haderslev
  - Research Site, Hillerød, Hillerod
  - Research Site, Middelfart, Middelfart
  - Research Site, Rønde, Ronde
  - Research Site, Tønder, Tonder

REFERENCES:
- [Derived] Emborg C, Hallerback T, Jorgensen L, Carlborg A. A retrospective study of clinical usage of quetiapine XR and quetiapine IR in outpatients with schizophrenia in Denmark. Hum Psychopharmacol. 2012 Sep;27(5):492-8. doi: 10.1002/hup.2254. PMID 22996616